CLINICAL TRIAL: NCT07314359
Title: Rapid Effects of a Biofield Patch on Antioxidant Status and Cellular Energy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 206-003
Record Dates: First submitted 2025-11-30; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Antioxidant Status
Keywords: Superoxide dismutase activity; Glutathione; Mitochondria; Cytokines

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, cross-over study design, followed by a 1-week open-label phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Crossover group 1, randomized (Experimental): Participants wear an active biofield patch versus a placebo patch for 12 hours on each of the two clinic days, at least 1 week apart, allowing for 1 week wash-out period between each patch. The order of interventions for this group is A, B. Following the blinded phase there will be an open-label phase where participants wear the active patch each day for 1 week until the final clinic visit.
  Interventions: Other: Active dermal patch; Other: Placebo dermal patch
- Experimental: Crossover group 2, randomized (Experimental): Participants wear a placebo patch versus an active biofield patch for 12 hours on each of the two clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. The order of interventions for this group is B, A. Following the blinded phase there will be an open-label phase where participants wear the patch each day for 1 week until the final clinic visit.
  Interventions: Other: Active dermal patch; Other: Placebo dermal patch

INTERVENTIONS:
Other: Active dermal patch — Non-transdermal patch
Other: Placebo dermal patch — Non-transdermal patch

SUMMARY:
The goal for this clinical proof-of-concept study is to compare an active biofield skin patch to a placebo patch on antioxidant function and mitochondrial function. A double-blind, placebo-controlled cross-over study design will be used.

DETAILED DESCRIPTION:
The goal for this clinical proof-of-concept study is to document acute effects of a photobiomodulating non-transdermal patch compared to a placebo patch, in an acute randomized double-blind placebo-controlled cross-over design. An add-on open-label module involves wearing the active patch daily for a week before the final clinic visit.

Data on endogenous antioxidant protection will be collected. The testing will show whether wearing the patch leads to a change in antioxidant activity of superoxide dismutase and glutathione. Data on cellular energy production and mitochondrial resilience in white blood cells under oxidative and inflammatory stress ex vivo will be collected. This testing will show whether using the active patch leads to changes in mitochondrial biogenesis and mitochondrial energy production under normal versus ex vivo-stressed conditions. Data on serum cytokine levels in both serum and serum-derived extracellular vesicles will be collected. The testing will show whether wearing the patch contributes to rapid change in pro- and anti-inflammatory markers and restorative growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18 - 75 years (inclusive);
* BMI between 18.0 and 34.9 (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with study procedures, including:

  * Maintaining a consistent diet and lifestyle routine throughout the study,
  * Consistent habit of bland breakfasts on days of clinic visits,
  * Abstaining from exercising and nutritional supplements on the morning of a study visit,
  * Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
  * Abstaining from music, candy, gum, computer/cell phone use (airplane mode is allowed), during clinic visits.

Exclusion Criteria:

* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Currently taking prescription weight loss drugs (such as semaglutide);
* Currently taking cholesterol-lowering medication (for example: statins);
* Currently experiencing intense stressful events/life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking anxiolytic, hypnotic, or anti-depressant prescription medication;
* Immunization during past 6 months;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Pregnant, nursing, or trying to become pregnant;
* Known allergies related to adhesive materials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Antioxidant protection | Baseline, 1 hour, and 2 hours after applying a patch.
  Data will be collected on intracellular levels of reduced glutathione and serum superoxide dismutase activity.

SECONDARY OUTCOMES:
Mitochondrial volume per cell | Baseline, 1 hour, and 2 hours after applying a patch.
  Mitochondrial volume per cell, measured by flow cytometry where the mean fluorescence intensity (MFI) is quantified on lymphocytes, monocytes, and polymorphonuclear cells. White blood cells are purified and cultured ex vivo in unstressed versus inflamed culture conditions. The mitochondrial reporter dye MitoTracker is used to obtain relative measures of mitochondrial volume per cell.
Mitochondrial membrane potential per cell | Baseline, 1 hour, and 2 hours after applying a patch
  Cellular energy production as a function of the mitochondrial membrane potential where the mean fluorescence intensity (MFI) is quantified on lymphocytes, monocytes, and polymorphonuclear cells. White blood cells are purified and cultured ex vivo in unstressed versus inflamed culture conditions. The mitochondrial reporter dye JC-1 is a fluorescent cationic dye used to obtain relative measures of mitochondrial membrane potential per cell.

OTHER OUTCOMES:
Communication in the body via serum cytokines | Baseline, 1 hour, and 2 hours after applying a patch.
  Data on serum levels of 27 pro- and anti-inflammatory cytokines and regenerative growth factors will be collected.
Communication in the body via cytokines in extracellular vesicles | Baseline, 1 hour, and 2 hours after applying a patch.
  Data on the levels of 27 pro- and anti-inflammatory cytokines and regenerative growth factors in serum extracellular vesicles will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No